CLINICAL TRIAL: NCT02012621
Title: Quantifying Drug Adherence and Drug Exposure to Antiretroviral Therapy.
Acronym: 2104
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 13-2104
Record Dates: First submitted 2013-12-04; First posted 2013-12-16 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-10

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; Adherence; Tenofovir; Dried Blood Spots
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate cumulative exposure to tenofovir diphosphate (TFV-DP) using dried blood spots (DBS) in treated HIV-infected patients who are receiving a TFV-based regimen. Using DBS will allow the investigators to assess this simple method to measure drug exposure in the clinical setting. The investigators hypothesize that TFV-DP levels will be lowest in individuals with a detectable viral load and highest in those with viral suppression.

DETAILED DESCRIPTION:
Antiretroviral drug exposure is directly linked to individual host factors which include age, weight, diet, and genetics. However, the main factor impacting long-term drug exposure is drug adherence. Adherence is a strong predictor of HIV treatment outcomes, but measuring adherence is difficult due to the inaccuracy of self-reporting and other commonly used monitoring methods. To date, no gold standard measure to monitor antiretroviral exposure and adherence has been applied in clinical practice. Tenofovir (TFV) and its active metabolite, tenofovir diphosphate (TFV-DP), have distinctive pharmacological characteristics that make them ideal candidates for drug adherence and exposure monitoring. The long half life (~14-17 days) of TFV-DP in red blood cells (RBC) are properties well suited for monitoring average dose exposure over time. Based on these, the investigators propose that RBC levels of TFV-DP are an accurate and precise measure of long-term drug exposure in HIV-infected individuals. In addition, the investigators aim to quantify TFV-DP in dried blood spots (DBS) as a simple method to measure drug exposure.

This is an observational, 48-week prospective study of HIV-infected individuals treated with TFV in which the investigators will compare DBS TFV-DP levels in virologically suppressed vs. non-suppressed individuals and evaluate the utility of TFV-DP in DBS to predict virologic failure and also drug toxicity. To accomplish this, the investigators will approach HIV-infected patients currently taking TFV (which is being prescribed by a primary care physician) and who present to the clinic for regular HIV care. After informed consent is obtained, the investigators will collect extra blood samples for DBS TFV-DP and obtain information on drug adherence. The investigators will also collect extra blood samples for DBS TFV-DP at each subject's subsequent visit for approximately 3 visits in a 48 week period of time.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected individual.
* 18 years and older.
* Taking tenofovir.
* Blood drawn during regular clinic visit.

Exclusion Criteria:

* Refusal to participate.
* Pregnancy.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected individuals who are taking tenofovir.
Sampling Method: Non-Probability Sample
Enrollment: 807 (Actual)
Dates: Start 2013-12; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose R. Castillo-Mancilla, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado-Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Derived] Morrow M, MaWhinney S, Coyle RP, Coleman SS, Gardner EM, Zheng JH, Ellison L, Bushman LR, Kiser JJ, Anderson PL, Castillo-Mancilla JR. Predictive Value of Tenofovir Diphosphate in Dried Blood Spots for Future Viremia in Persons Living With HIV. J Infect Dis. 2019 Jul 19;220(4):635-642. doi: 10.1093/infdis/jiz144. PMID 30942881
- [Derived] Castillo-Mancilla JR, Morrow M, Coyle RP, Coleman SS, Gardner EM, Zheng JH, Ellison L, Bushman LR, Kiser JJ, Mawhinney S, Anderson PL. Tenofovir Diphosphate in Dried Blood Spots Is Strongly Associated With Viral Suppression in Individuals With Human Immunodeficiency Virus Infections. Clin Infect Dis. 2019 Apr 8;68(8):1335-1342. doi: 10.1093/cid/ciy708. PMID 30137238
- [Derived] Castillo-Mancilla J, Seifert S, Campbell K, Coleman S, McAllister K, Zheng JH, Gardner EM, Liu A, Glidden DV, Grant R, Hosek S, Wilson CM, Bushman LR, MaWhinney S, Anderson PL. Emtricitabine-Triphosphate in Dried Blood Spots as a Marker of Recent Dosing. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6692-6697. doi: 10.1128/AAC.01017-16. Print 2016 Nov. PMID 27572401

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Cohort: 807 persons living with HIV (PLWH) on tenofovir disoproxil fumarate (TDF) at baseline were followed for up to three visits or 48 weeks.
Period: Overall Study
Arm/Group | Study Cohort
Started | 807
Visit 1 Completed | 807
Visit 2 Completed | 688
Visit 3 Completed | 444
Completed | 807
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: TFV-DP concentrations in DBS were available from 532 participants over three visits or 48 weeks. TFV-DP concentrations in DBS were available from 521 participants at baseline. Demographics from the full cohort (N=807) are reported here.
Arm/Group | Study Cohort
Number analyzed (Participants) | 807
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [37 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126
  Male | 681
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black | 149
  Race/Ethnicity: White | 472
  Race/Ethnicity: Hispanic | 147
  Race/Ethnicity: Other | 39

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Odds Ratio of Level of Tenofovir-diphosphate (TFV-DP) in Dried Blood Spots (DBS) Associated With Odds of HIV Viral Suppression at All Study Visits
Description: HIV viral load, binary cutoff at assay level of detection (<20 copies/mL vs. >= 20 copies/mL); reference group: drug concentration (TFV-DP) < 350 femtomole (fmol)/punch vs. drug concentration (TFV-DP) >= 1850 fmol/punch; adjusted odds ratio calculated using generalized estimating equations; concentration cutoffs established in prior research of healthy volunteers
Time Frame: Up to 48 Weeks
Population: Drug concentrations were available from 532 participants
Measure: Number (95% Confidence Interval); unit: Adjusted odds ratio (aOR)
Arm/Group | Study Cohort
Number analyzed (Participants) | 532
Adjusted odds ratio (aOR) | 73.5 [25.7 to 210.5]
Statistical Analysis 1: Comparison: Study Cohort; Test type: Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 73.5, 95% CI 2-sided [25.7 to 210.5]

2. Primary Outcome: Adjusted Odds Ratio of Three-month Self-reported Adeherence Associated With Odds of HIV Viral Suppression at All Study Visits
Description: HIV viral load, binary cutoff at assay level of detection (<20 copies/mL vs. >= 20 copies/mL); reference group: three-month self-reported adherence <28.5% vs. three-month self-reported adherence 100%; adherence cutoffs established in prior research
Time Frame: Up to 48 Weeks
Population: Three-month self-reported adherence data were available from 482 participants
Measure: Number (95% Confidence Interval); unit: Adjusted odds ratio (aOR)
Arm/Group | Study Cohort
Number analyzed (Participants) | 482
Adjusted odds ratio (aOR) | 8.5 [2.3 to 30.9]
Statistical Analysis 1: Comparison: Study Cohort; Test type: Other; p = 0.0012, Regression, Logistic; Odds Ratio (OR) = 8.5, 95% CI 2-sided [2.3 to 30.9]

3. Primary Outcome: Adjusted Odds Ratio of Level of Tenofovir-diphosphate (TFV-DP) in Dried Blood Spots (DBS) Associated With Odds of HIV Viral Suppression at Next Study Visit
Description: HIV viral load, binary cutoff at assay level of detection (<20 copies/mL vs. >= 20 copies/mL); drug concentration (TFV-DP) <800 femtomole (fmol)/punch) vs reference group of drug concentration (TFV-DP) >= 1650 fmol/punch; adjusted odds ratio calculated using generalized estimating equations
Time Frame: Up to 48 Weeks
Population: Paired drug concentration (TFV-DP) and HIV VL assessments were available from 451 participants
Measure: Number (95% Confidence Interval); unit: Adjusted odds ratio (aOR)
Arm/Group | Study Cohort
Number analyzed (Participants) | 451
Adjusted odds ratio (aOR) | 4.7 [2.6 to 8.7]
Statistical Analysis 1: Comparison: Study Cohort; Test type: Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.7, 95% CI 2-sided [2.6 to 8.7]

ADVERSE EVENTS:
Time Frame: N/A: observational study where samples were collected at the time of normally scheduled clinic visits
Description: N/A: observational study where samples were collected at the time of normally scheduled clinic visits; AEs not assessed
Arm/Group | Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT02012621/Prot_SAP_000.pdf